CLINICAL TRIAL: NCT03149692
Title: Penile Allograft Transplantation for Men With Penile Loss After Ritual Circumcision
Brief Title: Penile Transplant Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Andre van der Merwe, Associate Professor, University of Stellenbosch
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: N11/07/243
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Penile Amputation

STUDY DESIGN:
Intervention Model Description: Proof of concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penile allograft (Experimental): Penile human allografts transplanted
  Interventions: Other: Penile allograft transplantation

INTERVENTIONS:
Other: Penile allograft transplantation — Proof of concept of surgical procedure

SUMMARY:
One case of unsuccessful penile transplantation has been reported from China. The patient had suffered an industrial machine accident and lost his penis to the level of the pubic skin. Unfortunately the patient's wife insisted at about two weeks post-operatively that the organ be removed. At the time of surgical removal the penis was viable, except for a degree of superficial skin necrolysis. This has sparked debate on ethical issues regarding penile transplantation. South Africa is uniquely positioned in Sub-Saharan Africa and worldwide with relatively advanced medical services and a high prevalence of ritual circumcision practice with reports of high morbidity and mortality in the last 20 years. The substantial number of young men left with a severe penile defect or complete loss of the penis [9] creates a possible place for penile allograft transplantation as a treatment option.

DETAILED DESCRIPTION:
Literature review and rationale Ritual circumcision has been practised for centuries in Africa and other parts of the world. Clinical trials have shown that adult male circumcision, if performed correctly, could play a role in the prevention of HIV transmission and protect against invasive penile cancer. The prevalence of ritual circumcision practiced in Eastern and Southern Africa varies from about 80% in Kenya to about 20% in Uganda and Southern Africa. The procedure referred to as ritual circumcision is performed in a non-clinical environment by a traditional circumcisionist with no formal medical training. The main geographical area for this rite of passage in South Africa is among the Xhosa-speaking people of the Eastern Cape.

The complications of this procedure may lead to severe genital mutilation with partial or complete penile loss and may even result in mortality. In a study by Meissner and Buso conducted in the Eastern Cape from 2001 to 2005 there were 1748 hospital admissions, 107 genital mutilations and 177 deaths caused by ritual circumcision. Septicaemia, pneumonia and dehydration were the most common causes of death. The extent of genital mutilation varied from partial loss of the glans or distal penile shaft and urethra, to complete loss of the penis due to gangrene. Less common complications of ritual circumcision include polyarticular septic arthritis. The complication rates of ritual circumcision are much higher than those reported for infant and neonatal circumcision (1-7%) where the complications are mostly minor and almost never result in penile loss However, in a systematic review of the literature Wilcken et al found that the acquisition of data from the ritual circumcision studies was often poor, as only 11 of 1639 articles reviewed were suitable for analysis. Other causes of penile loss include electrical burns, self-mutilation and shotgun wounds. These aetiologies are rare in South Africa in contrast to the large numbers of ritual circumcision related penile amputees.

Figure 2. Loss of penis after a ritual circumcision complication and a ventilated critically ill patient with a septic penis after ritual circumcision. (Own pictures) The current treatment for total penile loss is surgical total penile reconstruction (TPR), also called total phallus reconstruction. The goal of TPR is to create a cosmetically acceptable, sensate penis, functional urethra that extends up to the distal glans which permits voiding in a standing position, and providing enough bulk to allow the insertion of a penile prosthesis for sexual intercourse. In addition, the donor-site should cause minimal morbidity and should be easy to conceal. The above goals are difficult to obtain in South African state patients, as penile prostheses are not available due to their high cost (about ZAR 80 000 per inflatable prosthesis).

The most widely used TPR technique is a radial forearm free flap (RFFF) described by Song et al in 1982. However the urethrocutaneous fistula rate is up to 40% and the donor site morbidity around 9%. The tissue flap is taken from the inside of the forearm and the defect covered with a skin graft. The flap is fashioned into the shape of a penis and a skin tube created inside to connect to the urethra. This flap may contain radial bone to provide rigidity and enable sexual function. Radial bone harvesting increases the morbidity of the donor site, as the forearm becomes very thin distally. The operation takes around 7 - 10 hours to perform. It provides a phallus which is cosmetically acceptable after tattooing the glans penis, but completely incapable of sexual function without a prosthesis, if bone is not incorporated. In a series of 15 adult female to male gender reassignment patients, only 7 received prostheses, indicating that not all TPRs are suitable to receive a prosthesis.

An artificial penile prosthesis is expensive and not available to state patients in SA due to lack of funding. These prostheses can extrude (especially with repeated sexual intercourse) or become infected. Jarow et al found 21.7% risk of infection if a penile reconstructive procedure was done with prostheses surgery. Infection of prostheses normally necessitates removal.

Other less commonly used types of tissue flaps for TPR are:

1. Free osteocutaneous fibula flap described by Sadove et al in 1993 with significant donor site and urethral complications of strictures (32%) and fistulas (16 %).
2. Free scapular flap described by Rorich et al in 1997, which has been reported in limited patient numbers.
3. Vertical rectus abdominis flap described by Santi et al in 1988.
4. Suprapubic abdominal wall flap reported by Bettocchi et al in 85 patients who underwent gender re-assignment, with urethral complications in 75%.

It is clear from the above that free flap TRP has many difficulties. The fact that several techniques have been described indicates that a single satisfactory operation with acceptable outcomes does not exist.

Most of the reported series were comprised of patients with gender dysphoria. Men requiring TPR for penile loss after ritual circumcision differ radically from most cases in the literature, in that these young men were subjected to a life-threatening event, often under peer pressure. Apart from the physical disfigurement, there is severe psychosocial debilitation resulting from the loss of sexual function and fertility. The reality in South African state hospitals is that the operative time and resources to provide free flap TPR for these patients is rarely available. If such surgery is performed, it is rarely followed by prosthesis placement, due to the high cost and the risk of complications such as extrusion and infection. Consequently, many mutilated young men face a future with severe sexual and psychosocial problems.

Transplantation of human body structures other than organs such as the heart, liver, pancreas and kidney is known as composite tissue allotransplantation (CTA) and has been practised for years in centres with available expertise. In 1998 Dubernard et al transplanted a forearm harvested from a brain dead man to 48-year old man. By 2009 at least 40 hand transplants had been performed, with very few immunological rejections and minimal immunosuppressive treatment in many cases . A possible explanation of this immune tolerance is that a type of chimerism is achieved, possibly due to the presence of bone marrow in the graft.

Allograft cadaver penis transplantation as treatment for penile loss from ritual circumcision could have the following benefits:

1. Psychological improvement
2. Cosmetic improvement
3. Sexual function re-established
4. Penile sensation re-established
5. Fertility restored
6. Shorter operation time

The negative factors are the following:

1. Immunosuppressive therapy to prevent organ rejection, which may be long-term
2. Intensive and comprehensive pre-operative counselling of the recipient and his spouse or partner
3. The necessity for long-term follow-up. One case of penis transplantation has been described in a man who lost his penis in an industrial machine accident. The donor was a young brain-dead male whose parents consented to the procedure. The Ethics review board of the hospital approved the procedure, which took 5 hours to perform. The penis survived 14 days and was viable, but the wife of the recipient then insisted that the penis be removed. At the time of amputation the corpora cavernosa and corpus spongiosum were viable. However, the skin suffered from superficial epidermal necrolysis that was diagnosed histologically. Venous congestion was evident on the penile skin, but no mention was made of anastomosis of the superficial dorsal vein of the penis.

Zhang et al debated the ethical issues of penis transplantation and expressed concerns about the body image expectations of the recipient and the fact that a cadaver would be buried without a penis. He concluded that good communication with the donor family would be essential. Dubernard (who performed the first hand transplant) commented on the single penis transplantation case and stressed that it is experimental but feasible. He expressed concern that the skin may be highly immunogenic and may be rejected separately from the rest of the penis. He also said that hand and face transplantation used to be a myth and a dream and has now turned into a reality.

ELIGIBILITY:
Inclusion Criteria:

* Male patients 18 years or older with total or partial penile loss as a complication from ritual circumcision, who are willing and able to provide written, informed consent.

Exclusion Criteria:

* Immunosuppression (HIV positive, diabetes mellitus or drugs affecting immune response) Active tuberculosis (TB) or a history of TB Previous forearm free flap Disorders of circulation (e.g. peripheral vascular disease, vasculitis) History of prior malignancy Renal failure and not on a renal replacement programme Systemic disease deemed by the investigator serious enough to preclude the use of immunosuppression agents Mental illness Patients who are unwilling, unable or unlikely to comply with immunosuppressive treatment and regular follow-up.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Must be males with loss of penis after ritual circumcision
Enrollment: 2 (Actual)
Dates: Start 2011-11-11 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Urinary function | 3 months after surgery
  Normal standing urination (subjects/patients had to sit to urinate before)
Sexual function | 3 months
  Normal sexual intercourse as for the subject - with or without medication assistance measured with IIEF score
Quality of life score | 6 months post operative
  Improved (or not) measured QoL with SF 36 software

CONTACTS AND LOCATIONS:
Overall Officials: Rafique Moosa, PhD, Study Director — University Stellenbosch
Locations (1):
- Stellenbosch University - Faculty of Medicine and Health Sciences, Division Urology, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Via publication or request. Low subject numbers expected